CLINICAL TRIAL: NCT02441894
Title: Cabazitaxel in Combination With Prednisolone With Primary Prophylaxis With PEG-G-CSF for the Treatment of Patients With Metastatic Castration-Resistant Prostate Cancer
Brief Title: Combination of Cabazitaxel With Prednisolone With Primary Prophylaxis With PEG-G-CSF in Treatment of Patients With Prostate Cancer
Acronym: PEGAZUS
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Sanofi (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CABAZL07239; U1111-1155-8055 (UTN)
Record Dates: First submitted 2015-05-08; First posted 2015-05-12 (Estimated); Last update posted 2017-01-24 (Estimated); Status verified 2017-01

CONDITIONS: Prostate Cancer
MeSH Terms: conditions — Prostatic Neoplasms | interventions — cabazitaxel; pegylated granulocyte colony-stimulating factor, human; Prednisolone; dexchlorpheniramine; Diphenhydramine; Ranitidine; Metoclopramide; Granisetron; Ondansetron; Dexamethasone

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Cabazitaxel (Experimental): 25 mg/m^2 of cabazitaxel is given intravenously in combination with prednisolone 10 mg orally per day. PEG-G-CSF is administered subcutaneously 24 hours after the completion of cabazitaxel infusion once every 3 weeks.
  Antihistamine (dexchlorpheniramine or diphenhydramine), corticosteroids (dexamethasone), and H2 antagonist (ranitidine) premedications will be administered by IV infusion at least 30 minutes prior to each dose of cabazitaxel. A prophylactic antiemetic treatment (metoclopramide, granisetron, or ondansetron) should be given to the patients in all cycles.
  Interventions: Drug: CABAZITAXEL XRP6258; Drug: PEG-G-CSF; Drug: Prednisolone; Drug: Dexchlorpheniramine or Diphenhydramine; Drug: Ranitidine; Drug: Metoclopramide, Granisetron, or Ondansetron; Drug: Dexamethasone

INTERVENTIONS:
Drug: CABAZITAXEL XRP6258 — Pharmaceutical form:solution Route of administration: intravenous
  Other Names: JEVTANA
Drug: PEG-G-CSF — Pharmaceutical form:solution Route of administration: subcutaneous
  Other Names: G-LASTA
Drug: Prednisolone — Pharmaceutical form:tablet Route of administration: oral
Drug: Dexchlorpheniramine or Diphenhydramine — Pharmaceutical form:tablet, powder, or solution Route of administration: oral, intravenous or intramuscular
Drug: Ranitidine — Pharmaceutical form:tablet or solution Route of administration: oral, intravenous or intramuscular
Drug: Metoclopramide, Granisetron, or Ondansetron — Pharmaceutical form:tablet, powder, jelly, or solution Route of administration: oral, intravenous or intramuscular
Drug: Dexamethasone — Pharmaceutical form:tablet, capsule, or solution Route of administration: oral or intravenous

SUMMARY:
Primary Objective:

To assess the tolerability of cabazitaxel 25 mg per body surface area (m^2) with primary prophylactic polyethylene glycol-granulocyte-colony stimulating factor (PEG-G-CSF) in terms of the incidence rate of febrile neutropenia (FN) (defined: absolute neutrophil count [ANC] <1000 per volume [mm^3] and a single temperature of >38.3 degree or a sustained temperature of ≥38 degree Celsius for more than one hour) during Cycle 1.

Secondary Objective:

To assess overall rate of FN and grade ≥3 neutropenia and diarrhea; frequencies of dose delay due to adverse events (AEs); dose reduction due to AEs; relative dose intensity; incidences of FN-related hospitalization and use of intravenous (IV) anti-infectives; tolerability according to National Cancer Institute Common Terminology Criteria for Adverse Events (NCI-CTCAE) v4.0; prostate specific antigen (PSA) response (50% decrease); tumor response according to Response Evaluation Criteria in Solid Tumors (RECIST) v1.1 if available.

DETAILED DESCRIPTION:
The total duration of study is 254 days as maximum with 14 days for screening, maximum of 21 days times 10 cycles for treatment, and 30 days for follow up.

ELIGIBILITY:
Inclusion criteria:

* Patients with metastatic castration-resistant prostate cancer (mCRPC) previously treated with chemotherapy including docetaxel.
* Male patients.
* Patients must have either measurable or nonmeasurable disease, or documented rising PSA levels.
* Patients signed informed consent.

Exclusion criteria:

* Age <20 at registration.
* Eastern Cooperative Oncology Group (ECOG) performance status (PS) ≥2.
* Inadequate organ and bone marrow function at registration as evidenced by:

  * Hemoglobin <10.0 g/dL.
  * ANC <5 x 10^9/L.
  * Platelet count <100 x 10^9/L.
  * Aspartate transaminase (AST) and/or alanine aminotransferase (ALT) >1.5 x upper limit of normal (ULN).
  * Total bilirubin >1.0 x ULN.
  * Serum creatinine >1.5 x ULN. Serum creatinine is 1.0-1.5 x ULN and creatinine clearance is under 60 mL/min (calculated according to Chronic Kidney Disease Epidemiology Collaboration [CKD-EP]).
* Prior isotope therapy or radiotherapy to ≥30% of bone marrow. At the first study drug administration day, patient has not elapsed 8 weeks (12 weeks for strontium-89) from the day prior isotope therapy finished.
* Prior surgery, radiation, chemotherapy, or other anticancer therapy within 4 weeks prior to enrollment in the study.
* Symptomatic peripheral neuropathy grade ≥2 (NCI CTCAE v.4.0).
* History of severe hypersensitivity reaction (grade ≥3) to polysorbate 80 containing drugs.
* Prior and other concurrent malignancy, excepted cases are as follows; basal cell carcinoma or squamous cell carcinoma of skin, or superficial (pTis, pTa, and pT1) bladder cancer (including immunotherapy) treated adequately, any other cancer completed the chemotherapy more than 5 years ago and been more than 5 years as disease free duration.
* Uncontrolled severe illness or medical condition (including uncontrolled diabetes mellitus).
* Known lesion at brain or leptomeninx.
* Known acquired immunodeficiency syndrome (AIDS-related illnesses) or known human immunodeficiency virus (HIV) disease requiring antiretroviral treatment.
* Active varicella zoster infection, anti-hepatitis C virus (HCV) antibody-positive (excluding patients negative for HCV virus in blood test or non-active seropositive patients with no hepatic abnormalities [AST, ALT, etc.]), or hepatitis B surface (HBs) antigen-positive.
* Concurrent or planned treatment with strong inhibitors or strong inducers of cytochrome P450 3A4 or 5 (wash-out period for a one week is necessary for patients who are already on these treatments or a two-week wash-out period is necessary for patients who are already on these treatments).
* Contraindication to be used corticosteroid.
* Patients with reproductive potential who do not agree to use an accepted and effective method of contraception during the study treatment period. The definition of "effective method of contraception" will be based on the Investigator's judgment.
* Participation in another clinical trial and any concurrent treatment with any investigational drug within 30 days prior to registration.
* Prior history of severe hypersensitivity reaction (≥grade 3) or intolerance to prednisolone, PEG-G-CSF or G-CSF.
* Known hypersensitivity to the component of PEG-G-CSF and/or G-CSF.
* Myelogenous leukemia insufficient decrease of the number of blast in bone marrow, or found myeloblast in peripheral blood.

The above information is not intended to contain all considerations relevant to a patient's potential participation in a clinical trial.

Min Age: 20 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 21 (Actual)
Dates: Start 2015-04; Primary Completion 2016-02 (Actual); Study Completion 2016-11 (Actual)

PRIMARY OUTCOMES:
Number of patients with FN (all grades) during study Cycle 1 | 3 weeks (during study Cycle 1)

SECONDARY OUTCOMES:
Number of patients with FN (all grades) | Up to 7 months as treatment period
Number of patients with Grade ≥3 neutropenia | Up to 7 months as treatment period
Number of patients with Grade ≥3 diarrhea | Up to 7 months as treatment period
Number of dose delays in the start of drug administration due to AEs | Up to 7 months as treatment period
Number of dose reductions due to AEs | Up to 7 months as treatment period
Percent change in relative dose intensity due to AEs | Up to 7 months as treatment period
Number of patients with FN-related hospitalization | Up to 7 months as treatment period
Number of patients who used IV anti-infective drugs | Up to 7 months as treatment period
Changes of PSA levels from baseline | Up to 7 months as treatment period
Number of patients with adverse events | Up to 7 months as treatment period

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Sciences & Operations, Study Director — Sanofi
Locations (8):
- Japan (8):
  - Investigational Site Number 392004, Chuo-ku, Chiba
  - Investigational Site Number 392008, Kita-gun
  - Investigational Site Number 392007, Kobe-shi, Hyogo
  - Investigational Site Number 392005, Nagakute-shi, Aichi
  - Investigational Site Number 392006, Osaka Sayama-shi, Osaka
  - Investigational Site Number 392001, Shinjuku-ku, Tokyo
  - Investigational Site Number 392009, Yokohama
  - Investigational Site Number 392002, Yokohama-shi, Kanagawa

REFERENCES:
- [Derived] Kosaka T, Uemura H, Sumitomo M, Harada K, Sugimoto M, Hayashi N, Yoshimura K, Fukasawa S, Ecstein-Fraisse E, Sunaga Y, Oya M. Impact of pegfilgrastim as primary prophylaxis for metastatic castration-resistant prostate cancer patients undergoing cabazitaxel treatment: an open-label study in Japan. Jpn J Clin Oncol. 2019 Aug 1;49(8):766-771. doi: 10.1093/jjco/hyz051. PMID 31329922